CLINICAL TRIAL: NCT01182935
Title: Elevated Triglyceride Levels and Later Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Tromso (Other)
Responsible Party: Rolf Jorde, Univesity of Tromsø
Other Study IDs: UIT-ENDO-2010-3
Record Dates: First submitted 2010-08-11; First posted 2010-08-17 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Type 2 Diabetes
Keywords: vitamin D; triglycerides; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- participants in the 4th Tromsø study

SUMMARY:
Subjects with elevated serum triglycerides in the 4th Tromso study in 1994/1995 were re-examined with an oral glucose tolerance test to see predictive value of triglycerides regarding development of type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* participants in the 4 Tromso study 1994 and with elevated serum triglyceride levels

Exclusion Criteria:

* type 2 diabetes

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: participants in the 4 Tromsø study 1994 and with elevated serum triglyceride levels
Sampling Method: Non-Probability Sample
Enrollment: 3509 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects with type 2 diabetes diagnosed with oral glucose tolerance test (OGTT) | At study enrollment in 2010

SECONDARY OUTCOMES:
The relation between serum 25(OH)D levels and blood glucose levels at OGTT | At study enrollment in 2010

CONTACTS AND LOCATIONS:
Overall Officials: rolf jorde, md, Principal Investigator — University of Tromso
Locations (1):
- Univesity of Tromsø, Tromsø, Tromsø, Norway